CLINICAL TRIAL: NCT00430586
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Multicenter Trial to Determine the Optimal Dose of NT 201, Free of Complexing Proteins, in the Treatment of Glabellar Frown Lines
Brief Title: Finding of Optimal Dose for NT 201 in the Treatment of Glabellar Frown Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Public Disclosure Manager, Merz Pharmaceuticals GmbH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MRZ 60201-0527/1
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- 20 U NT 201 (Experimental)
  Interventions: Drug: Botulinum neurotoxin type A, free of complexing proteins
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 10 U NT 201 (Experimental)
  Interventions: Drug: Botulinum neurotoxin type A, free of complexing proteins
- 30 U NT 201 (Experimental)
  Interventions: Drug: Botulinum neurotoxin type A, free of complexing proteins

INTERVENTIONS:
Drug: Botulinum neurotoxin type A, free of complexing proteins — Single treatment with 10, 20 or 30 Units of NT 201 given as intramuscular treatment injections of equal amount to 5 sites on Day 0. The same volume of reconstituted study medication (0.6 mL per subject) was administered irrespective of the treatment group. The total dose volume was administered in equal aliquots to the 5 injection sites. Thus, each of the 5 injection sites was injected with 0.12 mL study medication per injection site.
  Other Names: BTX-A,; BoNT/A,; incobotulinumtoxinA (Xeomin)
  Arms: 10 U NT 201; 20 U NT 201; 30 U NT 201
Drug: Placebo — Single treatment with Placebo given as intramuscular treatment injections of equal amount to 5 sites on Day 0. A volume of reconstituted 0.6 mL per subject was administered. The total dose volume was administered in equal aliquots to the 5 injection sites. Thus, each of the 5 injection sites was injected with 0.12 mL Placebo per injection site.
  Arms: Placebo

SUMMARY:
NT 201 is a botulinum toxin type A preparation free of complexing proteins, i.e. free of proteins other than the active toxin. Injected into the muscle, NT 201 causes local weakening to full paralysis depending on the administered dose. Botulinum toxin type A is widely used for aesthetic treatment of facial lines. This study will determine the optimal dose of NT 201 in the treatment of glabellar frown lines.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe glabellar frown lines

Exclusion Criteria:

* Previous insertion of permanent material in the glabellar area
* Neuromuscular function disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2006-11; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Percentage of responders at maximum frown at Day 30 as assessed by the investigator according to Facial Wrinkle Scale (FWS) | Baseline (Day 0) to Day 30
  Responders on the FWS are defined as subjects with glabellar line severity of none (0) or mild (1).
  The Primary Analysis Set (PAS) will be used for all confirmatory tests for the primary efficacy variables of the co-primary endpoint. The PAS will consist of all subjects in the Full Analysis Set who have available assessments by the investigator for severity of glabellar frown lines at maximum frown on Day 30, as well as patient's assessment at Day 0 and Day 30. All analyses for this population will therefore use the same sample for both primary endpoints.
Percentage of responders at maximum frown at Day 30 as assessed by patient's assessment according to 4-point scale | Baseline (Day 0) to Day 30
  Responders will be subjects with at least a 1-point improvement compared to Day 0.
  The Primary Analysis Set (PAS) will be used for all confirmatory tests for the primary efficacy variables of the co-primary endpoint. The PAS will consist of all subjects in the Full Analysis Set who have available assessments by the investigator for severity of glabellar frown lines at maximum frown on Day 30, as well as patient's assessment at Day 0 and Day 30. All analyses for this population will therefore use the same sample for both primary endpoints.

SECONDARY OUTCOMES:
Percentage of responders at maximum frown at Day 90 as assessed by the investigator according to FWS | Baseline (Day 0) to Day 90
  Responders on the FWS are defined as subjects with glabellar line severity of none (0) or mild (1).
  Secondary efficacy endpoints will be analyzed analogously to the analysis of primary efficacy endpoint.
Percentage of responders at maximum frown at Day 90 as assessed by patient's assessment | Baseline (Day 0) to Day 90
  Responders will be subjects with at least a 1-point improvement compared to Day 0.
  Secondary efficacy endpoints will be analyzed analogously to the analysis of primary efficacy endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Merz Pharmaceuticals, Study Chair — Merz Pharmaceuticals GmbH
Locations (1):
- Merz Pharmaceuticals GmbH, Frankfurt, Germany